CLINICAL TRIAL: NCT06449053
Title: Preventing Iatrogenic Dependence Linked to Hospitalisation in Elderly Patients Hospitalised in Acute Geriatrics
Acronym: TAKE CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP (URCPSL)
Record Dates: First submitted 2024-05-23; First posted 2024-06-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: An Acute Pathology
MeSH Terms: interventions — Organizations

STUDY DESIGN:
Intervention Model Description: * Use of a dedicated e-health application. In order to promote the implementation of DILH prevention measures, we will use an e-health application developed specifically for the study by PRESAGE in the areas where the intervention will take place. This innovative application will be used on admission for all patients included in the acute geriatric sectors in which the intervention will be deployed. It will first assess the risk of DILH individually for each of the 6 risk factors, and then scale the risk for the patient. Once the risk assessment has been carried out, the system will immediately produce a document setting out the personalized care plan for each patient, and disseminate knowledge through documents aimed at patients and caregivers.
  * The use of portable, connected treadmills (Ezygain, CE marked)
  * The installation of motion detector lighting in hospital rooms
Masking Description: soins usuels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAKE CARE (Experimental): * Use of a dedicated e-health application. In order to promote the implementation of DILH prevention measures, we will use an e-health application developed specifically for the study by PRESAGE in the areas where the intervention will take place. This innovative application will be used on admission for all patients included in the acute geriatric sectors in which the intervention will be deployed. It will first assess the risk of DILH individually for each of the 6 risk factors, and then scale the risk for the patient. Once the risk assessment has been carried out, the system will immediately produce a document setting out the personalized care plan for each patient, and disseminate knowledge through documents aimed at patients and caregivers.
  * The use of portable, connected treadmills (Ezygain, CE marked)
  * The installation of motion detector lighting in hospital rooms
  Interventions: Procedure: ORGANIZATIONAL
- CURRENT CARE (No Intervention): soins usuels

INTERVENTIONS:
Procedure: ORGANIZATIONAL — A. a formalization of the recommendations to be applied to prevent DILH B. implemented and facilitated by an e-health application C. and will be based on adapting the hospital environment (connected mats, movement sensors, prescription assistance) D. and the dissemination of knowledge (production of summary and empowerment documents).
  Arms: TAKE CARE

SUMMARY:
Iatrogenic dependence linked to hospitalisation DILH is very frequent, severe but avoidable in 80% of cases. Extensive research has identified 6 main causes of DILH in the elderly, which interact and have common risk factors: immobilisation, falls, undernutrition, de novo urinary incontinence, confusion and drug side-effects.

Our main hypothesis is that promoting access to, knowledge of and implementation of good practice recommendations by healthcare staff (medical and paramedical) concerning DILH in the elderly, based on graded interventions and targeting the 6 main causes of DILH, via the TAKE CARE intervention could reduce the incidence of DILH in the population of patients aged 75 or over hospitalised in acute geriatric units excluding post-operative and post-resuscitation, in the context of unscheduled hospitalizations.

A Multicenter, randomized, cluster trial evaluating the effect of the TAKE CARE intervention compared with usual care in patients will be conducted across 11 acute geriatric services in France. A total of 2200 patients will be needed for a total period of 6 months with a 6 months followup prior inclusion. Data will be collected directly from the patients' medical records and entered by an investigator or a clinical study technician in an electronic CRF (CleanWeb) managed by the URC PSL.

The trial will also include a qualitative component to assess, among other things, the implementation aspects of this complex intervention (individual interviews, focus group). A medico-economic component with a cost-utility analysis to assess the incremental cost-utility ratio, and a hospital microcosting study to assess the costs associated with the TAKE CARE intervention.

The impact of the TAKE CARE intervention will be studied using a "win-ratio" approach based on a hierarchical composite criterion that takes into account vital status at D7 and the change in ADL score between D15 before admission and D7. The difference in ADL score between D-15 and D7 will be compared between the 2 randomisation groups using a mixed linear model with the randomisation arm as a fixed effect and a random effect on the cluster. A win-ratio significantly greater than 1 will allow us to conclude that the TAKE CARE intervention is effective.

DETAILED DESCRIPTION:
Hospitalization for an acute illness in older individuals is connected to a decline in functionality, referred to as iatrogenic dependence linked to hospitalization (DILH). This is characterized by the inability to perform essential daily activities necessary for independent living. The literature has identified six primary causes of DILH in the elderly, which interact and share common risk factors. These causes include immobilization, falls, undernutrition, de novo urinary incontinence, confusion, and drug side effects. DILH is a prevalent issue, affecting approximately 40% of elderly patients admitted to the hospital. However, it is important to note that 80% of these cases can be prevented with appropriate measures.

Our primary hypothesis revolves around the idea that by promoting access to, knowledge of, and implementation of best practice recommendations among healthcare staff (both medical and paramedical) regarding DILH in the elderly, we can effectively reduce the incidence of DILH in the population of patients aged 75 or over who are hospitalized in acute geriatric units (excluding post-operative and post-resuscitation cases) during unscheduled hospitalizations. This will be achieved through the implementation of the TAKE CARE intervention, which is a multifaceted organizational intervention designed to facilitate the adoption of all current recommendations for combating DILH in the elderly, utilizing innovative equipment such as portable and connected treadmills, installation of lighting with motion detectors in hospital room and use of the SYNAPSEMed application .

A randomized, cluster trial will be conducted across 11 acute geriatric services in France to evaluate the impact of the TAKE CARE intervention compared to usual care in patients. The trial will span over a period of 6 months, during which a total of 2200 patients will be included. Half of the patients (n=1,100) will be admitted to the 11 wings of the geriatric ward in the INTERVENTION arm, while the other half (n=1,100) will be assigned to the 11 wings in the control arm. Following the inclusion period, the patients will be followup for a period of 6 months. Demographic and clinical data will be collected from the patients' medical records and entered into an electronic CRF (CleanWeb) by either an investigator or a clinical study technician. The URC PSL will manage the CRF through the eTAKE-CARE® application, as well as the SynapseMed® application. Data management and statistical analysis will be conducted by the PSL-CFX URC, using either the statistical software R version 3.6.3 or later (R Foundation for Statistical Computing, Vienna, Austria, https://www.R-project.org/) or SAS (SAS Institute Inc., Cary, NC, USA).

The trial will also include a qualitative component to assess, among other things, the implementation aspects of this complex intervention (individual interviews, focus group). A medico-economic component with a cost-utility analysis to assess the incremental cost-utility ratio, and a hospital microcosting study to assess the costs associated with the TAKE CARE intervention. QALYs (quality of life) will be assessed using the EQ5D-3L scale, which is robust in the geriatric population. Two aspects will be taken into account when estimating the cost utility, one will be the costs attributable to the purchase and immobilisation of the equipment necessary for the implementation of the intervention, and on the other hand, the costs associated with operating this equipment in relation to patient care.

The effectiveness of the TAKE CARE intervention will be examined through the utilization of a "win-ratio" method, which employs a hierarchical composite criterion. This criterion considers the vital status at D7 and the change in ADL score between D15 prior to admission and D7. By comparing the difference in ADL score between D-15 and D7 in the two randomization groups using a mixed linear model, with the randomization arm as a fixed effect and a random effect on the cluster. A win-ratio significantly greater than 1 will allow us to conclude that the TAKE CARE intervention is effective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 ans
* Unscheduled hospitalisation in one of the participating departments for an acute pathology, excluding post-operative care

Exclusion Criteria:

* Patients with a usual ADL score (assessed 15 days before hospitalisation) of 0
* Stay > 72 hours in another facility before admission to UGA
* Opposition to participation in the study (trusted support person / guardian - curator)
* Not affiliated to a social security scheme (beneficiary or beneficiary entitled)
* Patient under AME

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DILH will be assessed by the difference in ADL score between the pre-admission state and the ADL score at D7 | Through study time period, an average of 16 months
  DILH will be assessed by the difference in the ADL score (Activities of Daily Living Independence Scale) between the pre-admission state (assessment on admission of the ADL score under usual living conditions corresponding to the ADL score 15 days before hospitalisation, as it is usually measured in the acute geriatric ward), and the ADL score on Day 7 (7th day of hospitalisation).

SECONDARY OUTCOMES:
The change in ADL score between pre-admission status and J 7, as well as the change in ADL score between pre-admission status and hospital discharge, between admission and J 7, between pre-admission status and M3 and M6 | Through study time period, an average of 16 months
  The change in ADL score between pre-admission status and J 7
DILH will also be assessed by a new autonomy score currently under development to measure the effect of the intervention on each of the risk factors | Through study time period, an average of 16 monthes
  DILH will also be assessed by a new autonomy score currently

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.